CLINICAL TRIAL: NCT05568693
Title: Sequential Enhanced Safety Study of a Novel Coronavirus mRNA Vaccine in Adults Aged 18 Years and Older Who Have Completed 3 Doses of a New Inactivated Coronavirus Vaccine.
Brief Title: Sequential Enhanced Safety Study of a Novel Coronavirus Messenger RNA (mRNA) Vaccine in Adults Aged 18 Years and Older.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Yu Qin (Other)
Responsible Party: Sponsor-Investigator, Yu Qin, Director Technician, West China Second University Hospital
Organization: West China Second University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022069
Record Dates: First submitted 2022-09-30; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Corona Virus Disease 2019(COVID-19)
Keywords: COVID-19; Vaccine; mRNA; Safety; Immunogenicity; >=18 years; 3 doses of Inactivated COVID-19 vaccine
MeSH Terms: conditions — COVID-19 | interventions — mRNA Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mRNA-enhanced immunoem (Experimental): 1 dose of 0.3 ml of mRNA vaccine
  Interventions: Biological: 0.3ml of mRNA vaccine

INTERVENTIONS:
Biological: 0.3ml of mRNA vaccine — Subjects received 0.3ml of mRNA vaccine intramuscularly

SUMMARY:
This trial is a clinical study to evaluate the safety of sequential boosters of novel coronavirus mRNA vaccine in adults aged 18 years and older who have completed three doses of novel inactivated coronavirus vaccination. According to the results of the previous phase I clinical trial, the incidence of adverse reactions in the 0.3 ml dose group was lower than that in the 0.5 ml dose group, and the degree of adverse reactions was weaker. The dose of 0.3ml was chosen for the current study, and a 1-dose immunization program was completed for safety observation.

DETAILED DESCRIPTION:
According to the results of the preliminary phase I clinical trial, the incidence of adverse reactions in subjects in the 0.3 ml dose group was lower than in the 0.5 ml dose group and the degree of adverse reactions was weaker. The dose of 0.3ml was chosen for the current study.

The trial was designed to enroll 800 adult subjects aged 18 years and older who had completed three doses of inactivated New Coronavirus vaccine with an interval of more than 6 months between doses, and the proportion of elderly people aged 60 years and older was approximately 20%. Subjects will receive 0.3 ml of mRNA vaccine, complete a 1-dose immunization program, and undergo safety observations.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above adults.
* Able and willing to comply with the requirements of the clinical trial protocol and able to sign the informed consent form.
* Willing to discuss medical history with the investigator or physician and allow access to all medical records related to this trial.

Subjects have completed 3 doses of inactivated vaccine with at least 6 months between the last dose.

Exclusion Criteria:

* Subject is unfit to participate in the study based on the investigator's judgment.
* History of Middle East Respiratory Syndrome (MERS), Severe Acute Respiratory Syndrome(SARS) or other coronavirus infection or disease or history of related immunizations.
* Prior history of severe allergic reactions or hypersensitivity to vaccines or drugs, such as urticaria, severe skin eczema, dyspnea, laryngeal edema, hemangioma, etc., or history of serious adverse reactions associated with vaccines and/or history of severe anaphylactic reactions (e.g., systemic allergic reactions) to any component of the study vaccine.
* Immunocompromised individuals with known or suspected immunodeficiency as determined by medical history and/or physical examination, inability to control autoimmune disease, etc.
* Bleeding constitutional or condition associated with prolonged bleeding, which the investigator believes is contraindicated by intramuscular injection.
* Positive urine pregnancy test or lactating women, volunteers or their partners who have plans to become pregnant within 6 months.
* Severe hypertension and uncontrolled by medication (at the time of field measurement: systolic blood pressure ≥ 160 mmHg and diastolic blood pressure ≥ 100 mmHg).
* Suffering from a serious chronic disease or in a progressive stage that cannot be controlled smoothly, such as severe diabetes mellitus, thyroid disease, etc.
* Previously suffering from serious cardiac diseases such as myocarditis and pericarditis.
* Those who have planned to receive other vaccines within 28 days before or after the trial vaccination.
* Those receiving immunosuppressive therapy, including cytotoxic drugs or systemic corticosteroids, such as treatment for cancer or autoimmune disease, or are scheduled to receive treatment throughout the study period. If systemic corticosteroids are used for a short period of time (<14 days) for the treatment of an acute disease, subjects should not be allowed to enter this study until at least 28 days after corticosteroid therapy has ceased prior to study vaccination. Inhalation/spray, intra-articular, intra-bone, or topical (skin or eye) corticosteroid use is permitted.
* Have received or plan to receive blood/plasma products or immunoglobulins throughout the study period 60 days prior to study inoculation.
* Participated in other studies involving interventional studies within 28 days prior to study entry and/or during study participation.
* Have participated in other interventional studies involving lipid-containing nanoparticles.
* Have suspected COVID-19 symptoms such as respiratory symptoms, fever, cough, shortness of breath, and dyspnea.
* Axillary temperature >37.0°C or use of over-the-counter medications such as antipyretics and analgesics (e.g. acetaminophen, ibuprofen, naproxen, etc.) within 12 hours prior to experimental vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2023-03-21 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the incidence of adverse reactions (AR) in all subjects within 28 days of exemption | 28 days post vaccination
  Incidence of adverse reaction (AR)
Evaluation of the incidence of Serious Adverse Event (SAE) and Adverse Event of Special Interest (AESI) in all subjects at 6 months after exemption | 6 months post vaccination
  Incidence of Serious Adverse Event (SAE) and Adverse Event of Special Interest (AESI)

SECONDARY OUTCOMES:
Evaluation of the incidence of adverse reactions in all subjects at 30 minutes post-dispensing | 30 minutes post vaccination
  Incidence of adverse reaction (AR)
Evaluation of the incidence of adverse events in all subjects within 28 days of exemption | 28 days post vaccination
  Incidence of adverse events (AE)

CONTACTS AND LOCATIONS:
Locations (1):
- West China Second University Hospital, Chengdu, China